CLINICAL TRIAL: NCT02423655
Title: A Randomized, Controlled Trial to Evaluate Routine and Deferred Dialysis Initiation in Chinese Population
Brief Title: Routine and Deferred Dialysis Initiation
Acronym: RADDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Sichuan Academy of Medical Sciences (Other); First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other); Peking Union Medical College Hospital (Other); Shengjing Hospital (Other); The First Affiliated Hospital of BaoTou Medical College (Other); Beijing Hospital, National Center of Gerontology (Unknown); Beijing Haidian Hospital/Beijing Haidian Section of Peking University Third Hospital (Unknown); Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other); First Hospital of China Medical University (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li Zuo, Head of the Nephrology Department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201502010
Record Dates: First submitted 2015-04-10; First posted 2015-04-22 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Algorithms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deffered Dialysis Initiation (Experimental): Algorithm for deferred dialysis intervention:
  initiating dialysis in the absence of symptoms in patients with an eGFR of 5 ml/min /1.73 m2 or less
  Interventions: Other: Algorithm for deferred dialysis intervention
- Routine dialysis Initiation (Active Comparator): Algorithm for routine dialysis intervention:
  initiating dialysis in the absence of symptoms in patients with an eGFR of 7 ml/min /1.73 m2 (which is the average GFR for patients in Beijing to start dialysis )
  Interventions: Other: Algorithm for routine dialysis intervention

INTERVENTIONS:
Other: Algorithm for deferred dialysis intervention — Use combined indications to guide researchers to defer dialyzing progressive CKD patients. Asymptomatic patient will not start dialysis treatment until his eGFR becomes less than 5 ml/min/1.73m2. Or until 1. Patient's Kraemer index is >6 or with overt fluid overload after trying all conservative means（including appropriate medicines） 2. Patient's Subjective Global Assessment method (SGA) assessment is grade C 3. Patients have indications for emergency dialysis 4. Sever symptoms which cannot be relieved by conservative treatment
  Arms: Deffered Dialysis Initiation
Other: Algorithm for routine dialysis intervention — Use combined indications to guide researchers to initiate dialysis in progressive CKD patients routinely. Researchers will start dialysis treatment for a patient when his eGFR reaches 7 ml/min/1.73m2 in asymptomatic patients.
  Or patients have indications below: 1. Patient's Kraemer index is >6 or with overt fluid overload after trying all conservative means（including appropriate medicines） 2. Patient's SGA assessment is grade C 3. Patients have indications for emergency dialysis 4. Sever symptoms which cannot be relieved by conservative treatment
  Arms: Routine dialysis Initiation

SUMMARY:
This study evaluates the efficacy and safety of deferred dialysis initiation in Chinese population. 16 tertiary hospitals across China will be randomly assigned into routine and deferred dialysis groups.

DETAILED DESCRIPTION:
The timing for initiating dialysis for progressive chronic kidney disease (CKD) patients is an important issue yet is not well established. There is a strong trend to early dialysis initiation for end stage renal disease (ESRD) patients over the past decades. However, observational data found that early initiation seemed to produce no benefit but additional burden to patients and the health care system. The IDEAL study, the only randomized, controlled trial (RCT) on this issue, found that all-cause mortality, comorbidities and quality of life had no difference between early (glomerular filtration rate, GFR 10-14ml/min/1.73m2) and late (GFR 5-7ml/min/1.73m2) dialysis starters. However there was a big limitation in this study that the difference for average GFR between two groups (12 ml/min/1.73 m2 vs. 9.8 ml/min/1.73m2) was not so separate. Recently, the Canadian Society of Nephrology have released a clinical practice guideline on this issue. The guideline recommends an "intent-to-defer" approach for dialysis initiation and to initiate dialysis in the absence of symptoms in patients with an estimated GFR of 6 ml/min /1.73 m2 or less. In this guideline the specialists also express that the optimal management of patients with an estimated GFR of 6 ml/min per 1.73 m2 or less is based on limited data. There is a gap in knowledge. This research will further evaluate the efficacy and safety of deferred dialysis initiation and fill in this gap. In this study, algorithms will be adopted to determine the timing of dialysis initiation for both routine and deferred dialiysis groups, and the only difference in these two algorithms is the GFR level to initiate dialysis (7 Vs. <5 ml/min per 1.73 m2). The theory that blood access (arteriovenous fistulas) can be timely prepared according to the past GFR decline trajectory will also be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Nondialysis-dependent stable CKD stage 4-5 patients (eGFR>7ml/min /1.73 m2)
2. Willing to choose dialysis as his renal replacement therapy method
3. Heart function: grade I or II (NYHA Functional Classification)

Exclusion Criteria:

1. The life expectancy of patients is estimated to be short (due to causes other than kidney disease);
2. Acute infection occurred in one month;
3. Myocardial infarction, NYHA class IV or stroke events within 3 months;
4. Uncontrolled malignancy;
5. Active viral hepatitis;
6. Active rheumatic disease;
7. Pregnant women, women intending to conceive after enrollment or breastfeeding woman;
8. Planning to take kidney transplantation within the study period;
9. With indices of emergency dialysis;
10. eGFR less than 7 ml/min/1.73m2 in first visit;
11. Under other clinical studies which has an impact on this study;
12. Unable to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality: Proportion of patients who die from any cause | From date of enrollment until the end of study, assessed up to 3 years
  Proportion of patients who die from any cause during observation period.
Acute nonfatal cerebro-cardiovascular events before dialysis initiation | From date of enrollment until the date of dialysis initiation, or the date of death from any cause,or the end of study, whichever came first, assessed up to 3 year
  Proportion of patients who suffer from acute nonfatal cerebro-cardiovascular events before dialysis initiation.
  Cerebro-cardiovascular events include acute myocardial infarction,acute coronary ischemia syndrome,acute heart failure, acute exacerbation of chronic heart failure ,severe arrhythmia, stroke, etc.
Acute nonfatal cerebro-cardiovascular events after dialysis initiation | From date of dialysis initiation until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 year
  Proportion of patients who suffer from acute nonfatal cerebro-cardiovascular events after dialysis initiation.
  Cerebro-cardiovascular events include acute myocardial infarction,acute coronary ischemia syndrome,acute heart failure, acute exacerbation of chronic heart failure ,severe arrhythmia, stroke, etc.

SECONDARY OUTCOMES:
Hospitalization: Proportion of patients who are admitted to hospital | From date of enrollment until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 year
  Proportion of patients who are admitted to hospital
Nutrition assessment | From date of enrollment until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 years, performed every 3 months
  SGA assessment and serum albumin level are used to assess nutrition status
Patient reported outcome of quality of life | From date of enrollment until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 years, once every 3 months
  The short form health survey questionnaire 36 will be used.
Complications of dialysis | From date of dialysis initiation until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 year
  Proportion of patients who suffer from dialysis complications including blood acess infection, thrombosis, hypotension, etc.
Costs | From date of enrollment until the date of death from any cause,or the end of study, whichever came first, assessed up to 3 years, performed every 3 months
  All money patients and insurance agency spend on medical care related with CKD
Arteriovenous fistulas usage | From date of enrollment until the date of dialysis initiation, assessed up to 3 years
  Proportion of patients using arteriovenous fistulas as their blood access when dialysis initiation. The timing for preparing arteriovenous fistulas depends on the past GFR decline trajectory
Catheter usage | From date of enrollment until the date of dialysis initiation, assessed up to 3 years
  Proportion of patients using catheter as their blood access when dialysis initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Rosansky SJ, Cancarini G, Clark WF, Eggers P, Germaine M, Glassock R, Goldfarb DS, Harris D, Hwang SJ, Imperial EB, Johansen KL, Kalantar-Zadeh K, Moist LM, Rayner B, Steiner R, Zuo L. Dialysis initiation: what's the rush? Semin Dial. 2013 Nov-Dec;26(6):650-7. doi: 10.1111/sdi.12134. Epub 2013 Sep 19. PMID 24066675
- [Result] Cooper BA, Branley P, Bulfone L, Collins JF, Craig JC, Fraenkel MB, Harris A, Johnson DW, Kesselhut J, Li JJ, Luxton G, Pilmore A, Tiller DJ, Harris DC, Pollock CA; IDEAL Study. A randomized, controlled trial of early versus late initiation of dialysis. N Engl J Med. 2010 Aug 12;363(7):609-19. doi: 10.1056/NEJMoa1000552. Epub 2010 Jun 27. PMID 20581422
- [Result] Crews DC, Scialla JJ, Boulware LE, Navaneethan SD, Nally JV Jr, Liu X, Arrigain S, Schold JD, Ephraim PL, Jolly SE, Sozio SM, Michels WM, Miskulin DC, Tangri N, Shafi T, Wu AW, Bandeen-Roche K; DEcIDE Network Patient Outcomes in End Stage Renal Disease Study Investigators. Comparative effectiveness of early versus conventional timing of dialysis initiation in advanced CKD. Am J Kidney Dis. 2014 May;63(5):806-15. doi: 10.1053/j.ajkd.2013.12.010. Epub 2014 Feb 6. PMID 24508475
- [Result] Nesrallah GE, Mustafa RA, Clark WF, Bass A, Barnieh L, Hemmelgarn BR, Klarenbach S, Quinn RR, Hiremath S, Ravani P, Sood MM, Moist LM; Canadian Society of Nephrology. Canadian Society of Nephrology 2014 clinical practice guideline for timing the initiation of chronic dialysis. CMAJ. 2014 Feb 4;186(2):112-7. doi: 10.1503/cmaj.130363. No abstract available. PMID 24492525
- [Derived] Zhao X, Wang P, Wang L, Chen X, Huang W, Mao Y, Hu R, Cheng X, Wang C, Wang L, Zhang P, Li D, Wang Y, Ye W, Chen Y, Jia Q, Yan X, Zuo L. Protocol for a prospective, cluster randomized trial to evaluate routine and deferred dialysis initiation (RADDI) in Chinese population. BMC Nephrol. 2019 Dec 9;20(1):455. doi: 10.1186/s12882-019-1627-0. PMID 31818266
- See also: The website of Peking University People's Hospital — http://www.phbjmu.edu.cn/